CLINICAL TRIAL: NCT05834322
Title: Relationship Between Exercise, Physical Activity Levels, Sleep Quality and Cognitive Function Among Older Adults.
Brief Title: Exercise, PA, Sleep Quality and Cognitive Function Among Older Adults.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Changhua University of Education (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Lee, Graduate Student, National Changhua University of Education
Other Study IDs: NCUEREC-112-009
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Function
Keywords: physical activity; cognitive function; sleep; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rapid increase in the prevalence of dementia in Taiwan poses an economic burden on healthcare systems as well as the families of the patients. Thus, how to prevent dementia is a crucial issue. Mild cognitive impairment (MCI) is defined as cognitive decline objectively and subjectively and it has been deemed as a transitional state between normal cognition and dementia. Identifying and preventing MCI can be a venue for reducing the prevalence of dementia. Sleep and physical activity are modifiable risk factors of MCI. Both factors could influence brain structure, such as the volume of the hippocampus. As a result, physical activity and adequate sleep are helpful to prevent the decline of cognitive function. In addition, sleep could regulate physical activity and change cognitive function indirectly. To our knowledge, there has been no research investigating the relationship between sleep, physical activity, and cognitive function in Taiwan. Hence, this research will aim to explore the relationship between sleep, physical activity, and cognitive function. Whether sleep and physical activity can be predictors of MCI will be investigated. We will recruit 150 participants aged above 65, who haven't been diagnosed with MCI or dementia. The measurements will include the Chinese version of The Pittsburgh Sleep Quality Index (PSQI), the Chinese Version of the Physical Activity Scale for the Elderly (PASE-C), and the Chinese version of Montreal Cognitive Assessment (MoCA). The relationship between sleep, physical activity level, and cognitive function will be analyzed by multiple linear regression and Pearson correlations. A prediction equation will be established.

ELIGIBILITY:
Inclusion Criteria:

* aged above 65
* haven't been diagnosed with MCI or dementia
* be able to read and write in Chinese

Exclusion Criteria:

* elders who unable to talk or communicate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants should be over 65 and haven't been diagnosed with MCI or dementia.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | at the time the participants enroll
  Chinese version of Montreal Cognitive Assessment (MoCA) will be use to assess cognitive function
Sleep quality | at the time the participants enroll
  Chinese version of The Pittsburgh Sleep Quality Index (PSQI) will be use to assess sleep quality
Physical activity levels | at the time the participants enroll
  Chinese Version of the Physical Activity Scale for the Elderly (PASE-C) will be use to assess physical activity levels

CONTACTS AND LOCATIONS:
Locations (1):
- National Chunghua University of education, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided